CLINICAL TRIAL: NCT03992547
Title: The Effects of Gait Performance and Brain Activity After Robot-assisted Gait Training(RAGT) On Patients With Lower Extremity Thermal Injury : a Prospective, Randomized, Single-blinded Study
Brief Title: The Effects of Robot-assisted Gait Training(RAGT) On Patients With Burn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Translational Research Program for Rehabilitation Robots (NRCTR-EX19002) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HangangSHH-4
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-06

CONDITIONS: Burns
Keywords: funcional near infrared spectroscopy; Robot-assisted gait training
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- robot assisted gait traing (Experimental): SUBAR® (CRETEM, Korea) is a wearable robot with a footplate that assists patients to perform voluntary muscle movements. RAGT enables training of automatically programmed normal gait pattern. Patients underwent 30 min of RAGT using SUBAR® and conventional exercise rehabilitation each for 30 min once a day for 5 days a week for 12 weeks.
  Interventions: Other: Robot-assisted Gait Training

INTERVENTIONS:
Other: Robot-assisted Gait Training — SUBAR® (CRETEM, Korea) is a wearable robot with a footplate that assists patients to perform voluntary muscle movements. RAGT enables training of automatically programmed normal gait pattern.

SUMMARY:
This study aimed to elucidate the efficacy and investigate the mechanism of motor recovery after RAGT on patients with lower extremity burn. To investigate RAGT effects, we compare the results of RGAT group to the results of matched conventional(CON) rehabilitation group.

DETAILED DESCRIPTION:
Gait enables individuals to move forward and is considered a natural skill. However, gait disturbances are very common in patients with burn injury. Major causes of functional impairment are pain and joint contractures. Contractures at the lower extremities such as the hip, knee, and ankle significantly limit gait. Recent studies focused on the application of robot-assisted gait training (RAGT).

This single-blinded, randomized, controlled trial involved 40 patients with lower extremity burns. Patients were randomized into a RAGT or a CON group.

SUBAR® (CRETEM, Korea) is a wearable robot with a footplate that assists patients to perform voluntary muscle movements. RAGT enables training of automatically programmed normal gait pattern. Patients underwent 30 min of RAGT using SUBAR® and conventional exercise rehabilitation each for 30 min once a day for 5 days a week for 12 weeks. The CON group focused on gait training such as passive ROM exercise, weight bearing training, manual lymphatic drainage, and hypertrophic scar care for 60 min once a day for 5 days a week for 12 weeks.

A wearable functional near-infrared spectroscopy (fNIRS) device has been developed for studying cortical hemodynamics. Changes in cortical activity has not previously been documented in patients with burn injury. Cortical activity was measured by evaluating relative changes in oxyhemoglobin level. The NIRST Analysis Tool v2.1 was utilized to analyze fNIRS data in a MATLAB environment. Functional scores of functional ambulation category (FAC), 6-minute walking test (6MWT) distances, and numeric rating scale (NRS) scores of pain before and after 12 weeks RAGT were measured. Numeric rating scale (NRS) was used to rate the degree of subjective pain during gait movement: 0 points were assigned when no pain was noted, and unbearable pain was assigned 10 points. To evaluate functional recovery, FAC scores and 6-minute walking test (6MWT) distances were measured. FAC was evaluated based on six scales. Scale 0 means that the patient cannot walk or can only walk with assistance of two people. Scale 5 means that the patient can walk independently. We measured walking-related cortical activity using an fNIRS device before and after 12 weeks RAGT.

ELIGIBILITY:
Inclusion Criteria:

* the parients with lower extremity burn
* ≤1 functional ambulation category (FAC) score ≤ 3

Exclusion Criteria:

* cognitive disorders
* intellectual impairment before burn injury
* serious cardiac dysfunction
* problems with weight bearing due to unstable fractures
* body weight ≥100 kg
* severe fixed contracture
* skin disorders that could be worsened by robot assisted gait training

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2020-07-30 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Functional ambulation category (FAC) | 12 weeks intervention
  FAC was evaluated based on six scales. Scale 0 means that the patient cannot walk or can only walk with assistance of two people. Scale 5 means that the patient can walk independently.
6-minute walking test (6MWT) | 12 weeks intervention
  6MWT was performed in accordance with standardized guidelines, and the walking course was 20 m. Patients were instructed to walk as far as possible in 6 min
Numeric rating scale (NRS) scores | 12 weeks intervention
  Numeric rating scale (NRS) was used to rate the degree of subjective pain during gait movement: 0 points were assigned when no pain was noted, and unbearable pain was assigned 10 points.

SECONDARY OUTCOMES:
frontal lobe cortial activity | 12 weeks intervention
  A wearable functional near-infrared spectroscopy (fNIRS) device has been developed for studying cortical hemodynamics. Changes in cortical activity has not previously been documented in patients with burn injury. Cortical activity was measured by evaluating relative changes in oxyhemoglobin level. The NIRST Analysis Tool v2.1 was utilized to analyze fNIRS data in a MATLAB environment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeongdeungpo-Ku, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gawaziuk JP, Peters B, Logsetty S. Early ambulation after-grafting of lower extremity burns. Burns. 2018 Feb;44(1):183-187. doi: 10.1016/j.burns.2017.07.005. Epub 2017 Aug 5. PMID 28789801
- [Background] Bae YH, Ko YJ, Chang WH, Lee JH, Lee KB, Park YJ, Ha HG, Kim YH. Effects of Robot-assisted Gait Training Combined with Functional Electrical Stimulation on Recovery of Locomotor Mobility in Chronic Stroke Patients: A Randomized Controlled Trial. J Phys Ther Sci. 2014 Dec;26(12):1949-53. doi: 10.1589/jpts.26.1949. Epub 2014 Dec 25. PMID 25540505